CLINICAL TRIAL: NCT02076529
Title: A Study About Pharmacokinetic and Pharmacodynamics of Ramosetron in Chemotherapy Induced Nausea and Vomiting
Brief Title: Phamacokinetic and Pharmacodynamic Study of Ramosetron in Chemotherapy Induced Nasea and Vomiting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonnam National University Hospital (Other)
Responsible Party: Principal Investigator, Sang-Hee Cho, Assistant Professor, Chonnam National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: RamosetronPK
Record Dates: First submitted 2014-02-28; First posted 2014-03-03 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-02

CONDITIONS: Colon Cancer
Keywords: chemotherapy induced nausea vomiting
MeSH Terms: conditions — Colonic Neoplasms | interventions — ramosetron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ramosetron 0.6mg (Experimental): Ramosetron 0.6mg intravenous injection 30min before chemotherapy
  Interventions: Drug: Ramosetron 0.6mg
- Ramosetron 0.45mg (Experimental): Ramosetron 0.45mg intravenous injection 30min before chemotherapy
  Interventions: Drug: Ramosetron 0.45mg
- Ramosetron 0.3mg (Active Comparator): Ramosetron 0.3mg intravenous injection 30 min before chemotherapy
  Interventions: Drug: Ramosetron 0.3mg

INTERVENTIONS:
Drug: Ramosetron 0.3mg
  Other Names: Nasea 0.3mg
  Arms: Ramosetron 0.3mg
Drug: Ramosetron 0.45mg
  Other Names: Nasea 0.45mg
  Arms: Ramosetron 0.45mg
Drug: Ramosetron 0.6mg
  Other Names: Nasea 0.6mg
  Arms: Ramosetron 0.6mg

SUMMARY:
This study is designted to know optimal dose of Ramosteron to control for chemotherapy induced nasea and vomoting (CINV)based on its pharmacokinetics, pharmacodynamic study and clinilcal parameters using Rhodes Index.

DETAILED DESCRIPTION:
Nausea and vomiting is a common adverse event during chemotherapy treatment. Even if preventive medicines such as dopamine receptor antagonist, corticosteroid, serotonin receptor antagonist, has been developed and used, there is residual nausea and/or vomiting in a significant percentage of patients treated for cancer. Serotonin receptor antagonist is the most potent antiemetic agent and has been used widely. However, the optimal dose of serotonin antagnosit based on individual symptoms is not defined. Therefore, this study was conducted to design standardization model for optiomal serotonin antagonist concentration using pharmacodynamic study and Rhodes Index as a suggogate marker for CINV.

ELIGIBILITY:
Inclusion Criteria:

* Patients who recevied moderate emetogenic chemotherapy
* Age between 18-75
* ECOG PS 0-2
* Adequate organ fuction including bone marrow, liver and kidney

Exclusion Criteria:

* Gastrointestinal obstruction or carcinomatosis peritonei
* CNS metastasis or disability in CNS
* Intractable medical illness
* Pregnancy or inadequate contraception

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile of Ramosetron according to 3 level of dose | 10min to 48 hours post-dose
  Pharmacokinectics using NONMEM will be analyzed from serum after Ramosetron injection from 10 min to 48 hours (10min, 1hr, 6hr, 24hr, 48hr)

SECONDARY OUTCOMES:
Rhodes Index | 1 hour to seven days post-dose
  Monitor using Rhodes Index will be performed each time at 1hour, 6hour, 24hour, 48hour and seven dyas after Ramosetron injection

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Hee Cho, M.D.Ph.D., Principal Investigator — CNUHH
Locations (1):
- Chonnam National University Hwasun Hospital, Gwangju, Jeollanamdo, South Korea